CLINICAL TRIAL: NCT05410587
Title: Prospective First in Human Clinical Investigation to Evaluate the Safety of the Fracture Monitor T1 in Patients with Femur Fractures Treated with a Locking Compression Plate
Brief Title: Fracture Monitor - Femur
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: AO Innovation Translation Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FM_AO_001
Record Dates: First submitted 2022-04-28; First posted 2022-06-08 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Femoral Fracture
Keywords: Fracture fixation, internal; Femur; Fracture healing
MeSH Terms: conditions — Femoral Fractures

STUDY DESIGN:
Intervention Model Description: Multicenter prospective interventional clinical investigation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fracture Monitor T1 (implantable device class III) (Other)
  Interventions: Device: Fracture Monitor (implantable device class III)

INTERVENTIONS:
Device: Fracture Monitor (implantable device class III) — Femoral fracture fixation (bridge plating aiming at secondary bone healing) using a locking plate with an attached investigational Fracture Monitor T1.

SUMMARY:
Thirty-seven patients diagnosed with femoral fracture to be treated with a compatible plate will be enrolled for this multicenter prospective interventional study. The Fracture Monitor T1 will be attached to the locking plate during osteosynthesis. Prior to discharge, it will be connected to an app installed either on the patients' smartphone or on the smartphone provided by the sponsor. The device will continuously collect and process data, which can automatically be downloaded via Bluetooth through the smartphone app and transferred in encrypted form to a dedicated cloud server. The smartphones will be equipped with a basic app version with rudimentary user interface that has no data visualization function. During the rehabilitation phase, data collected by the device will not be accessible to the surgeon nor the patient to ensure that no therapeutic decision will be made based on the acquired data. Every patient is treated as per standard of care.

The primary objective of the study is to collect safety information of the Fracture Monitor T1. The secondary objectives are to collect information on device performance, device handling, and usability.

All adverse events (AEs) and serious AEs (SAEs) will be recorded during the study. These will be reviewed and evaluated for their potential relationship to the device.

All patients will be followed up for 6 months after the surgery according to the local standard of care. Given that the removal of the Fracture Monitor T1 may occur beyond 6 months, a safety follow-up will take place at the time point when the Fracture Monitor T1 is removed as per the instructions for use if it has not been removed within the 6 months.

The results will be compiled into a clinical evaluation report to be submitted as part of the technical documentation for the conformity assessment procedure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Closed growth plates at time of injury
* Femoral fracture requiring osteosynthesis and treated with one of the following plates:

  * DePuy Synthes LCP® 4.5/5, Broad
  * DePuy Synthes LCP® 4.5/5, Broad Curved
  * DePuy Synthes LCP® Condylar Plate 4.5/5.0
  * DePuy Synthes VA-LCP® Condylar Plate 4.5/5.0
  * DePuy Synthes LCP® Distal Femur
  * DePuy Synthes LCP® Proximal Femoral Plate 4.5/5.0
  * DePuy Synthes LCP® Proximal Femur Hook Plate
  * 41medical AG, Biphasic Plate DF
* ASA score 1-3
* Full weight-bearing capacity prior to the injury
* The patient is foreseen to be capable of postoperative weight bearing of at least 15 kg
* Willingness to undergo an additional surgery to remove the Fracture Monitor T1 if its removal is not done together with the fixation plate within two years according to standard of care
* Ability to provide written informed consent

Preoperative exclusion Criteria:

* Concomitant fractures in the contralateral leg
* Electromagnetic hypersensitivity
* Implanted electromagnetic bone stimulators
* Pregnancy (determined by pregnancy test)
* Prisoner
* Known history of substance abuse (eg, recreational drugs and alcohol) that would preclude reliable assessments
* Participation in any other medical device or medicinal product study within the previous month that could influence the results of the present clinical investigation

Intraoperative exclusion criteria:

* Use of compression lag screw across fracture fragment
* Compression osteosynthesis
* Precontouring of implant at the area of the attachment of Fracture Monitor T1
* Double-plating technique
* Soft-tissue coverage > 6 cm above the data logger
* Concurrent use of intramedullary nail
* Patients foreseen to require magnetic resonance imaging scanning at any part of the body or shockwave therapy at the proximity of the Fracture Monitor T1
* Fracture Monitor T1 not functional according to the instruction for use (IFU, section 24, A) and no functional replacement implant available

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Incidence of ADEs | 6 months postsurgery
  To evaluate the safety, (ie the incidence of adverse device effects (ADEs), of the investigational device Fracture Monitor T1 in femoral fracture patients)

SECONDARY OUTCOMES:
Clinical performance: Relationship - implant load/bone healing | 6 months
  Relationship between relative implant load and bone healing status
Clinical performance: Relationship - implant load/weight bearing | 6 months
  Relationship between relative implant load and prescribed weight bearing
Clinical performance: Relationship - implant load/Function Index for Trauma(FIX-IT) | 6 months
  Relationship between relative implant load and Function Index for Trauma (FIX-IT) score FIX-IT: max 12 points - 0 worse/12 best
Clinical performance: Relationship - implant load/Patient reported outcomes | 6 months
  Relationship between relative implant load and Patient reported outcomes: pain, EuroQol 5- dimension (EQ-5D) EQ-5D health states can be summarised using a 5-digit code or represented by a single summary number (index value) which reflects how good or bad a health state is according to the preferences of the general population of a country/region.
Clinical performance: Relationship - implant load/Modified Radiographic union score for tibia(mRUST) | 6 months
  Relationship between relative implant load and mRUST score. mRUST: The mRUST score ranges from 4-16 as the four cortices assessed in two orthogonal planes have a score range from 1 to 4 (1: absent callus - 4 callus remodeled)
Clinical performance: Curve drop | 6 months
  Analyses of the loading curve drop based on:
  -Time to curve drop
Clinical performance: Difference curve drop/soc x-ray | 6 months
  Analyses of the loading curve drop based on:
  * Difference in the timing between drop in the loading curve (50%) and standard-of-care x-ray
Other safety parameters: AEs | 6 months
  - Incidence of adverse events (AEs)
Other safety parameters: DD | 6 months
  - Incidence of device deficiencies within 6 months
Technical performance in a clinical setup | 6 months
  • Average minimum sensor strain per loading event
Technical performance in a clinical setup | 6 months
  • Daily active time of implant (patient activity triggers recording of implant)
Technical performance in a clinical setup | 6 months
  • Number of daily activations (implant switches from idle to recording)
Technical performance in a clinical setup | 6 months
  • User calibration range (patient-specific calibration on stiffness of fixation construct)
Technical performance in a clinical setup | 6 months
  • Data down and upload frequency
Technical performance in a clinical setup | 6 months
  • Number of Bluetooth adverts
Technical performance in a clinical setup | 6 months
  • Bluetooth signal strength (dBm)
Technical performance in a clinical setup | 6 months
  • Bluetooth connection time (s)
Technical performance in a clinical setup | 6 months
  • Battery voltage after each month
Technical performance in a clinical setup | 6 months
  • Power consumption (device lifetime)
Technical performance in a clinical setup | 6 months
  • Internal device temperature
Technical performance in a clinical setup | 6 months
  • Initialization and daily system test results
Technical performance in a clinical setup | 6 months
  • Internal clock accuracy

CONTACTS AND LOCATIONS:
Overall Officials: Benedikt Braun, Principal Investigator — University Hospital Tübingen
Locations (4):
- Germany (4):
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitätsklinikum Münster, Münster
  - Berufsgenossenschaftliche Unfallklinik Tübingen, Tübingen
  - Universitätsklinikum Ulm, Ulm

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Braun BJ, Raschke MJ, Schutze K, Pohlemann T, Joeris A, Ernst M. Prospective first-in-human clinical investigation to evaluate the safety of the fracture monitor T1 in patients with femur fractures treated with a locking compression plate: a study protocol. BMJ Open. 2025 Jul 30;15(7):e102749. doi: 10.1136/bmjopen-2025-102749. PMID 40744509